CLINICAL TRIAL: NCT03537599
Title: Phase I/II Clinical Trial of Daratumumab and Donor Lymphocyte Infusion in Patients With Relapsed Acute Myeloid Leukemia Post-Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Daratumumab and Donor Lymphocyte Infusion in Treating Participants With Relapsed Acute Myeloid Leukemia After Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor acccrual
Sponsor: Sumithira Vasu (Other)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17102; NCI-2018-00616 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Minimal Residual Disease; Recurrent Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Neoplasm, Residual; Leukemia, Myeloid, Acute | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DLI, daratumumab) (Experimental): Participants receive daratumumab intravenously once a week for 8 weeks and donor lymphocyte infusion in weeks 3 or 4 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Procedure: Donor Lymphocyte Infusion; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Procedure: Donor Lymphocyte Infusion — Given via infusion
  Other Names: DLI; Donor Leukocyte Infusion
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of donor lymphocyte infusions when given together with daratumumab and to see how well they work in treating participants with acute myeloid leukemia that has come back after a stem cell transplant. A donor lymphocyte infusion is a type of therapy in which lymphocytes (white blood cells) from the blood of a donor are given to a participant who has already received a stem cell transplant from the same donor. The donor lymphocytes may kill remaining cancer cells. Monoclonal antibodies, such as daratumumab, may interfere with the ability of cancer cells to grow and spread. Giving daratumumab and donor white blood cells may work better in treating participants with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety and tolerability of daratumumab and escalating doses of donor lymphocyte infusions (DLI) in post-hematopoietic cell transplantation (HCT) patients with relapsed acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) transformed to AML (phase I).

II. To evaluate overall response rate to daratumumab and DLI in patients with post-HCT relapsed AML and MDS (phase II).

SECONDARY OBJECTIVES:

I. To assess overall response rates in minimal residual disease (MRD) positive patients and in patients with overt morphological relapse.

II. To assess MRD conversion rates from MRD positive to MRD negative. III. To determine the post-relapse 6-month overall response (OS) rates of patients with relapsed AML and MDS following allogeneic hematopoietic stem cell transplantation (allo-HSCT) who are treated with daratumumab.

IV. To determine the rates of graft-versus-host disease (GVHD) (both grades II-IV and III-IV) and autoimmune side effects of daratumumab.

V. To determine the post-relapse 6-month progression-free survival (PFS) rates of patients with relapsed AML and MDS following allo-HSCT who are treated with daratumumab.

EXPLORATORY OBJECTIVES:

I. To compare CD38 expression levels in myeloid blasts and interferon gamma (IFN-y) levels in plasma at the time of relapse before starting daratumumab and at progression or relapse after daratumumab.

II. To compare peripheral blood T cell number and subsets (CD3, CD4, CD8, (CD38 expression on regulatory T cells [T-regs], CD4 and CD8), T regs, B-regulatory cells, natural killer (NK) cell numbers and bone marrow T cell subsets at the time of relapse before starting daratumumab, at the time of partial/complete response to daratumumab, and at the time of progression or relapse after daratumumab.

III. To evaluate whether daratumumab has (i) direct anti-leukemia effects (ii) antibody-dependent cellular cytotoxicity (ADCC) and antibody-dependent cellular phagocytosis (ADCP) and (III) immune modulation of autologous immune system (NK cells, T cells, T-regs, B-regulatory cells [B-regs], and myeloid-derived suppressor cells [MDSCS]) in AML.

IV. To evaluate the effect of daratumumab on exosome content and clearance along with other soluble factors in AML.

V. To evaluate serum interferon (IFN) levels pre-daratumumab, during and post-daratumumab.

VI. To evaluate whether fratricide occurs in patients treated with daratumumab.

OUTLINE: This is a phase I, dose escalation study of donor lymphocyte infusions followed by a phase II study.

Participants receive daratumumab intravenously once a week for 8 weeks and donor lymphocyte infusion in weeks 3 or 4 in the absence of disease progression or unacceptable toxicity. Participants found to be in complete response (CR) at the end of 8 weeks may receive daratumumab IV once every 2 weeks for 8 weeks, and then once monthly for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* AML relapse following Allo-HSCT (Morphological relapse, or MRD positive verified by flow cytometry, cytogenetics, and molecular mutations)
* Relapsed/Refractory AML must not be candidates for available therapies known to be effective for treatment of their AML.
* MDS transformed to AML following Allo-HCT
* Patients who received a 10/10 HLA-matched allogeneic HCT either from sibling donors or unrelated donors or atleast a 5/10 haploidentical transplant.
* Engraftment must have occurred as defined by platelet (PLT) count > 20,000/µL and ANC

  * 0.5
* Eastern Cooperative Oncology Group (ECOG) performance status < 3
* Creatinine clearance > 40 ml/min (calculated or measured)
* Aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN), alanine aminotransferase (ALT) < 3 x ULN
* Total bilirubin < 1.5 x ULN
* Off calcineurin inhibitors for at least 2 weeks
* Prednisone dose ≤ 20 mg/day
* Patients with proliferative disease can be cytoreduced with cytotoxic chemotherapy at Investigator discretion, but there should be at least a 14 day window between start of cytoreductive therapy and start of daratumumab
* Blast count ˂20K/day (hydrea use is allowed)

Exclusion Criteria:

* No demonstrable evidence of donor chimerism (˂ 55% donor CD3 or CD33 chimerism)
* Patients with a molecular mutation without chromosomal abnormalities or declining chimerisms (MRD status must be verified by surface marker and mutational analyses)
* Active graft-versus-host disease (GvHD) grades II-IV; prior acute GVHD could have occurred but resolved at time of initiation of daratumumab
* Extensive chronic GvHD requiring ongoing immunosuppression with calcineurin inhibitors
* Patients with FLT3+ AML or blast crisis CML who have not yet received post-transplant TKI therapy
* Active central nervous system (CNS) disease testicular disease

EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.; seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

* Patients must not have moderate or severe persistent asthma within the past 2 years and must not have currently uncontrolled asthma of any classification.
* History of grade IV anaphylactic reaction to monoclonal antibody therapy
* Active autoimmune disease prior to transplant
* Concurrent use of any other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to low enrollment dose levels were not increased during the study
Groups:
- Cohort I (High Risk AML); Cohort 2 (AML/MDS-relapsed After Allo-HSCT): Participants receive daratumumab intravenously once a week for 8 weeks and donor lymphocyte infusion in weeks 3 or 4 in the absence of disease progression or unacceptable toxicity.
  Daratumumab: Given IV
  Donor Lymphocyte Infusion: Given via infusion
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Cohort I (High Risk AML) | Cohort 2 (AML/MDS-relapsed After Allo-HSCT)
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Disease Progression | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (High Risk AML) | Cohort 2 (AML/MDS-relapsed After Allo-HSCT) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 70 [67 to 73] | 62.5 [58 to 67] | 66.25 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: patients]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility Defined as the Establishment of the Appropriate Dose Level of Donor Lymphocyte Infusion When Given With a Fixed Dose of Daratumumab
Time Frame: Up to 6 months
Population: Data was not collected due to participants not reaching time point
Arm/Group | Cohort I (High Risk AML) | Cohort 2 (AML/MDS-relapsed After Allo-HSCT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rates of Complete Remission
Description: Kaplan-Meier estimates of survival and relapse will be made. Response will be measured using standard criteria. For pre/post-treatment comparisons in the correlative part of the study, a paired t-test will be applied. Two-tailed p values <0.05 will be considered statistically significant in all analyses.
Time Frame: Up to 6 months
Population: Data was not collected due to participants not reaching time point
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Post-relapse Progression-free Survival
Description: as for outcome 2
Time Frame: At 6 months
Population: Data was not collected due to participants not reaching time point
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Post-relapse Overall Survival
Description: as for outcome 2
Time Frame: Up to 6 months
Population: Data was not collected due to participants not reaching time point
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Minimal Residual Disease (MRD) Conversion Rates
Time Frame: Up to 6 months
Population: Data was not collected due to participants not reaching time point
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Expression of CD38 on Bone Marrow
Description: CD38 expression on bone marrow is checked prior to transplant. Most patients are in remission prior to transplant. Patients who were initially treated at Ohio State University (OSU) will have banked leukemia samples at the time of diagnosis. Expression of CD38 on samples at diagnosis and prior to transplant by immunohistochemical staining will be performed.
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Expression of CD38 in Lymphocytes in Bone Marrow
Description: Percentage of lymphocytes in bone marrow pre- and post-treatment with daratumumab will be studied. In addition to percentage, expression of CD38 on lymphocytes will be evaluated by immunohistochemistry (IHC).
Time Frame: Baseline to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Phenotypic Studies to Evaluate T Cell Exhaustion/Function
Description: This will be performed on bone marrow samples pre-and post-treatment with Daratumumab at the specified time points.
Time Frame: Baseline to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Phenotypic Studies to Evaluate Activation Status of Natural Killer (NK) Cells
Description: This will be performed on bone marrow samples pre-and post-treatment with daratumumab.
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: T-cell, NK Cell, B-cell, and Myeloid-derived Suppressor Cells (MDSC) Infiltration in Bone Marrow
Description: This will be evaluated on bone marrow samples pre-and post-treatment with daratumumab.
Time Frame: Baseline to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Exosomes From Bone Marrow
Description: This will be examined for both number and also content (protein, messenger ribonucleic acid [mRNA], and micro RNAs [mIRs]).
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Serial Assessment of Microenvironment
Description: Will be assessed with with stromal cell cultures.
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Chimerism Analysis
Description: Using single-nucleotide polymorphisms, relative contributions from donor vs. recipient in sorted CD3+ and CD33+ cells will be measured and expressed as a percentage.
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Immune Reconstitution
Description: Dr.Gerard Lozanski has developed a panel called the Immunome to study reconstitution of T cells, NK cells and B cells post-transplant. Specific information regarding stages of activation of T cells is also available from this panel.
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Immune Response Post Daratumumab
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Phenotypic Studies to Evaluate T Cell Exhaustion
Description: This will be performed on bone marrow samples pre-and post-treatment with daratumumab.
Time Frame: Baseline to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Phenotypic Studies to Evaluate Activation Status of NK Cells
Description: This will be performed on bone marrow samples pre-and post-treatment with daratumumab.
Time Frame: Baseline to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

18. Other Pre Specified Outcome: Measurements of Cytokines Including But Not Limited to Interferon Gamma (IFN-y)
Description: This will be measured at relapse, pre and post daratumumab treatment. Exosomes from bone marrow will be examined at these serial times for both number and also content (protein, messenger ribonucleic acid [mRNA], and micro RNA [mIRs]).
Time Frame: Up to 6 months
Population: Not sufficient number of patients accrued to report on outcomes
Arm/Group | Treatment (DLI, Daratumumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected and monitored from the start of the study until study completion up to an average of 4 months.
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was used for grading patients adverse events.
Arm/Group | Cohort I (High Risk AML) | Cohort 2 (AML/MDS-relapsed After Allo-HSCT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (High Risk AML) (N=2) | Cohort 2 (AML/MDS-relapsed After Allo-HSCT) (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Bloody Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 1 (1) | 2 (6)
Fever (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (9) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Infusion related reaction (Immune system disorders) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (6) | 2 (3)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (7) | 2 (9)
Platelet count decreased (Investigations) | 2 (6) | 2 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (3) | 2 (9)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Folate Deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03537599/Prot_SAP_000.pdf